CLINICAL TRIAL: NCT04550312
Title: The Impact of Lifestyle Alteration by Strict Prevention Measures on Non-COVID Deaths in the Region With Low COVID-19 Transmission Rate
Brief Title: The Impact of Lifestyle Changes on Non-COVID Deaths
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2020-KL142-01
Record Dates: First submitted 2020-09-13; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Lifestyle Alteration; Non-COVID Deaths

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The increase of all-cause mortality in the areas with high COVID-19 transmission rate due to COVID-19 deaths and the collateral damage to other healthcare problems is well known. However, the COVID-19 mortality is very low in the regions with low transmission rate and sufficient medical resources. In such regions, strict prevention measures were taken and these would alter the people's lifestyle and hygienic habits and further impact on non-COVID-19 deaths. Yet, there has no thorough investigation in this aspect.

DETAILED DESCRIPTION:
Background The increase of all-cause mortality in the areas with high COVID-19 transmission rate due to COVID-19 deaths and the collateral damage to other healthcare problems is well known. However, the COVID-19 mortality is very low in the regions with low transmission rate and sufficient medical resources. In such regions, strict prevention measures were taken and these would alter the people's lifestyle and hygienic habits and further impact on non-COVID-19 deaths. Yet, there has no thorough investigation in this aspect.

Methods The number of registered deaths among 8.8 million permanent residents with specific causes from January 2018 to June 2020 were sourced from the Xuzhou Center for Disease Control and Prevention, Jiangsu Province, China. Death rates were calculated and compared by weeks, months, and years with a focus on the period of COVID-19 pandemic from Jan 24 to March 27, 2020. Numeric values of all-cause death and the death rates of non-COVID diseases were compared in time series at different time scales.

ELIGIBILITY:
Inclusion Criteria:

* All cases of death reported to the Xuzhou CDC during the study period

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all cases of non-Covid-19 deaths in Xuzhou region between 2018 and 2020
Sampling Method: Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Numeric values of all-cause death and the death rates of non-COVID diseases | from January 2018 to June 2020

CONTACTS AND LOCATIONS:
Overall Officials: minglong chen, PHD, Principal Investigator — Xuzhou Medical University affiliated hospital
Locations (1):
- Xuzhou Medical University affiliated Hospital, Xuzhou, Jiangsu, China